CLINICAL TRIAL: NCT02629887
Title: Non-inflatable Supraglottic Airway (NI-SGA) vs. Face Mask (FM) as a Primary Interface Device for Neonatal Resuscitation: A Pilot Study
Brief Title: Non-inflatable Supraglottic Airway (NI-SGA) vs. Face Mask (FM) as a Primary Interface Device for Neonatal Resuscitation
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study design changed for recruitment purposes; no participants enrolled
Sponsor: University of Oklahoma (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 5848
Record Dates: First submitted 2015-12-10; First posted 2015-12-14 (Estimated); Last update posted 2018-05-09 (Actual); Status verified 2018-05

CONDITIONS: Neonatal Resuscitation
Keywords: supraglottic airway; neonatal resuscitation; ventilation; term infant
MeSH Terms: conditions — Respiratory Aspiration | interventions — Masks

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Face Mask (Active Comparator): Standard Face Mask with T piece resuscitator for neonatal resuscitation. Face mask placement per Neonatal Resuscitation Program resuscitation guideline.
  Interventions: Device: Face Mask; Device: T-Piece Resuscitator
- Non-inflatable supraglottic airway (Active Comparator): Use of non-inflating supraglottic airway with T-piece resuscitator instead of Standard Face Mask with T piece resuscitator for neonatal resuscitation, replacing standard of care face mask in Neonatal Resuscitation Program guideline.
  Interventions: Device: Non-inflatable supraglottic airway; Device: T-Piece Resuscitator

INTERVENTIONS:
Device: Non-inflatable supraglottic airway — at delivery if resuscitation is required infant randomized to NI-SGA or face mask as the interface for positive pressure ventilation.
  Arms: Non-inflatable supraglottic airway
Device: Face Mask — at delivery - standard airway management per Neonatal Resuscitation Program utilizing face mask.
  Arms: Face Mask
Device: T-Piece Resuscitator — T-Piece Resuscitator for providing postivie pressure ventilation via face mask or non-inflatable supraglottic airway

SUMMARY:
Prospective, randomized controlled trial to be performed at one center, of term and late preterm infants requiring resuscitation. Prenatal consent will be obtained. At randomization, babies will be resuscitated following Neonatal Resuscitation Program (NRP) guidelines and ventilated using the T-piece resuscitator with either a Face Mask (FM) or Non-inflating supraglottic airway. Video will be collected during resuscitation as well as written documentation. Primary outcome will be time to spontaneous breathing, length of resuscitation, and need for endotracheal intubation.

DETAILED DESCRIPTION:
Mothers who are close to delivery of a term or near term infant with estimated fetal weight of 2500gms will be approached for consent to randomize their infant to resuscitation with mask or non-inflatable supraglottic airway (NISGA) if resuscitation is required. Study personnel in delivery will open sequential envelopes with randomized code to indicate which device is to be used if necessary. The resuscitator will be blinded until determination of need of respiratory support. At that time, the appropriate randomized device (face mask or NISGA) will be handed to the resuscitator for use along with T-Piece resuscitator. Video data capture will be used to record type, length and response to resuscitation. This information will be translated to a database prior to destruction of video.

ELIGIBILITY:
Inclusion Criteria:

* Newborns > or = 2000gms requiring positive pressure ventilation within the first 2 minutes of life

Exclusion Criteria:

* Newborns with expected fetal weight <2000 grams
* Known congenital malformations
* Multiple gestation (twins and above)
* History of meconium stained fluid

Max Age: 30 Minutes | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2018-04-15 (Estimated); Primary Completion 2018-04-15 (Estimated); Study Completion 2018-04-15 (Estimated)

PRIMARY OUTCOMES:
Time to Spontaneous Breathing | 30 minutes
  Record of time from beginning of resuscitation to time of spontaneous breathing
Duration of Positive Pressure Ventilation | 30 minutes
  Total time of positive pressure ventilation required to adequate spontaneous breathing.
Need for subsequent endotracheal intubation | 30 minutes
  Failure of non-invasive resuscitative efforts by face mask or NI-SGA requiring intubation per NRP guideline.

SECONDARY OUTCOMES:
Time needed for NI-SGA placement | 1 minute
  Time needed adequate placement of non-inflatable supraglottic airway
Need for drugs in resuscitation | 30 minutes
  Drug administration as part of the standard neonatal resuscitation per NRP
Use of Chest Compressions | 30 minutes
  Need for chest compressions as part of neonatal resuscitation per NRP guidelines
Use of oxygen | 30 minutes
  Amount and duration of oxygen use in resuscitation
Rate of complications associated with resuscitation | 30 minutes
  Presence of complications including bleeding, abdominal distension, laryngeal stridor
Heart rate 2 minutes after initiation of resuscitation | 2 minutes
  Heart rate assessed at 2 minutes
Maximum inspiratory pressure | 30 minutes
  Record of highest peak inspiratory pressure used in resuscitation

CONTACTS AND LOCATIONS:
Overall Officials: Arlen Foulks, DO, Principal Investigator — University of Oklahoma
Locations (1):
- University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Liu L, Oza S, Hogan D, Perin J, Rudan I, Lawn JE, Cousens S, Mathers C, Black RE. Global, regional, and national causes of child mortality in 2000-13, with projections to inform post-2015 priorities: an updated systematic analysis. Lancet. 2015 Jan 31;385(9966):430-40. doi: 10.1016/S0140-6736(14)61698-6. Epub 2014 Sep 30. PMID 25280870
- [Background] Ersdal HL, Singhal N. Resuscitation in resource-limited settings. Semin Fetal Neonatal Med. 2013 Dec;18(6):373-8. doi: 10.1016/j.siny.2013.07.001. Epub 2013 Jul 27. PMID 23896083
- [Background] Wyckoff MH, Perlman JM. Effective ventilation and temperature control are vital to outborn resuscitation. Prehosp Emerg Care. 2004 Apr-Jun;8(2):191-5. doi: 10.1016/j.prehos.2003.12.013. PMID 15060855
- [Background] Wyckoff MH, Perlman JM, Laptook AR. Use of volume expansion during delivery room resuscitation in near-term and term infants. Pediatrics. 2005 Apr;115(4):950-5. doi: 10.1542/peds.2004-0913. PMID 15805369
- [Background] Ersdal HL, Mduma E, Svensen E, Perlman JM. Early initiation of basic resuscitation interventions including face mask ventilation may reduce birth asphyxia related mortality in low-income countries: a prospective descriptive observational study. Resuscitation. 2012 Jul;83(7):869-73. doi: 10.1016/j.resuscitation.2011.12.011. Epub 2011 Dec 23. PMID 22198423
- [Background] Szyld E, Aguilar A, Musante GA, Vain N, Prudent L, Fabres J, Carlo WA; Delivery Room Ventilation Devices Trial Group. Comparison of devices for newborn ventilation in the delivery room. J Pediatr. 2014 Aug;165(2):234-239.e3. doi: 10.1016/j.jpeds.2014.02.035. Epub 2014 Mar 29. PMID 24690329
- [Background] Kattwinkel J, Perlman JM, Aziz K, Colby C, Fairchild K, Gallagher J, Hazinski MF, Halamek LP, Kumar P, Little G, McGowan JE, Nightengale B, Ramirez MM, Ringer S, Simon WM, Weiner GM, Wyckoff M, Zaichkin J; American Heart Association. Neonatal resuscitation: 2010 American Heart Association Guidelines for Cardiopulmonary Resuscitation and Emergency Cardiovascular Care. Pediatrics. 2010 Nov;126(5):e1400-13. doi: 10.1542/peds.2010-2972E. Epub 2010 Oct 18. No abstract available. PMID 20956432
- [Background] O'Donnell CP, Davis PG, Morley CJ. Positive pressure ventilation at neonatal resuscitation: review of equipment and international survey of practice. Acta Paediatr. 2004 May;93(5):583-8. doi: 10.1111/j.1651-2227.2004.tb02981.x. PMID 15174776
- [Background] Hartung JC, te Pas AB, Fischer H, Schmalisch G, Roehr CC. Leak during manual neonatal ventilation and its effect on the delivered pressures and volumes: an in vitro study. Neonatology. 2012;102(3):190-5. doi: 10.1159/000339325. Epub 2012 Jul 10. PMID 22796898
- [Background] Deindl P, O'Reilly M, Zoller K, Berger A, Pollak A, Schwindt J, Schmolzer GM. Influence of mask type and mask position on the effectiveness of bag-mask ventilation in a neonatal manikin. Eur J Pediatr. 2014 Jan;173(1):75-9. doi: 10.1007/s00431-013-2122-4. Epub 2013 Aug 11. PMID 23933670
- [Background] Schilleman K, van der Pot CJ, Hooper SB, Lopriore E, Walther FJ, te Pas AB. Evaluating manual inflations and breathing during mask ventilation in preterm infants at birth. J Pediatr. 2013 Mar;162(3):457-63. doi: 10.1016/j.jpeds.2012.09.036. Epub 2012 Oct 25. PMID 23102793
- [Background] Schmolzer GM, Kamlin OC, O'Donnell CP, Dawson JA, Morley CJ, Davis PG. Assessment of tidal volume and gas leak during mask ventilation of preterm infants in the delivery room. Arch Dis Child Fetal Neonatal Ed. 2010 Nov;95(6):F393-7. doi: 10.1136/adc.2009.174003. Epub 2010 Jun 14. PMID 20547584
- [Background] Foglia EE, Owen LS, Thio M, Ratcliffe SJ, Lista G, Te Pas A, Hummler H, Nadkarni V, Ades A, Posencheg M, Keszler M, Davis P, Kirpalani H. Sustained Aeration of Infant Lungs (SAIL) trial: study protocol for a randomized controlled trial. Trials. 2015 Mar 15;16:95. doi: 10.1186/s13063-015-0601-9. PMID 25872563
- [Background] Kattwinkel J, Perlman JM, Aziz K, Colby C, Fairchild K, Gallagher J, Hazinski MF, Halamek LP, Kumar P, Little G, McGowan JE, Nightengale B, Ramirez MM, Ringer S, Simon WM, Weiner GM, Wyckoff M, Zaichkin J. Part 15: neonatal resuscitation: 2010 American Heart Association Guidelines for Cardiopulmonary Resuscitation and Emergency Cardiovascular Care. Circulation. 2010 Nov 2;122(18 Suppl 3):S909-19. doi: 10.1161/CIRCULATIONAHA.110.971119. No abstract available. PMID 20956231
- [Background] Richmond S, Wyllie J. European Resuscitation Council Guidelines for Resuscitation 2010 Section 7. Resuscitation of babies at birth. Resuscitation. 2010 Oct;81(10):1389-99. doi: 10.1016/j.resuscitation.2010.08.018. No abstract available. PMID 20956046
- [Background] Schmolzer GM, Agarwal M, Kamlin CO, Davis PG. Supraglottic airway devices during neonatal resuscitation: an historical perspective, systematic review and meta-analysis of available clinical trials. Resuscitation. 2013 Jun;84(6):722-30. doi: 10.1016/j.resuscitation.2012.11.002. Epub 2012 Nov 9. PMID 23146881
- [Background] Leone TA, Rich W, Finer NN. A survey of delivery room resuscitation practices in the United States. Pediatrics. 2006 Feb;117(2):e164-75. doi: 10.1542/peds.2005-0936. PMID 16452326
- [Background] Schreiner MS, Feltman D, Wiswell T, Wootton S, Arnold C, Tyson J, Lantos JD. When is waiver of consent appropriate in a neonatal clinical trial? Pediatrics. 2014 Nov;134(5):1006-12. doi: 10.1542/peds.2014-0207. Epub 2014 Oct 6. PMID 25287456
- [Background] Nichol G, Huszti E. Design and implementation of resuscitation research: special challenges and potential solutions. Resuscitation. 2007 Jun;73(3):337-46. doi: 10.1016/j.resuscitation.2006.10.021. Epub 2007 Feb 9. PMID 17292525
- [Background] Paterson SJ, Byrne PJ, Molesky MG, Seal RF, Finucane BT. Neonatal resuscitation using the laryngeal mask airway. Anesthesiology. 1994 Jun;80(6):1248-53; discussion 27A. PMID 8010471
- [Background] Gandini D, Brimacombe JR. Neonatal resuscitation with the laryngeal mask airway in normal and low birth weight infants. Anesth Analg. 1999 Sep;89(3):642-3. doi: 10.1097/00000539-199909000-00018. No abstract available. PMID 10475295
- [Background] Zanardo V, Weiner G, Micaglio M, Doglioni N, Buzzacchero R, Trevisanuto D. Delivery room resuscitation of near-term infants: role of the laryngeal mask airway. Resuscitation. 2010 Mar;81(3):327-30. doi: 10.1016/j.resuscitation.2009.11.005. Epub 2009 Dec 22. PMID 20022416
- [Background] Zhu XY, Lin BC, Zhang QS, Ye HM, Yu RJ. A prospective evaluation of the efficacy of the laryngeal mask airway during neonatal resuscitation. Resuscitation. 2011 Nov;82(11):1405-9. doi: 10.1016/j.resuscitation.2011.06.010. Epub 2011 Jul 16. PMID 21763393
- [Background] Trevisanuto D, Cavallin F, Nguyen LN, Nguyen TV, Tran LD, Tran CD, Doglioni N, Micaglio M, Moccia L. Supreme Laryngeal Mask Airway versus Face Mask during Neonatal Resuscitation: A Randomized Controlled Trial. J Pediatr. 2015 Aug;167(2):286-91.e1. doi: 10.1016/j.jpeds.2015.04.051. Epub 2015 May 21. PMID 26003882
- [Background] Bernhard M, Benger JR. Airway management during cardiopulmonary resuscitation. Curr Opin Crit Care. 2015 Jun;21(3):183-7. doi: 10.1097/MCC.0000000000000201. PMID 25922892